CLINICAL TRIAL: NCT01902056
Title: Implant Placement and Simultaneous Soft Tissue Grafting With Single or Double Layers of Acellular Dermal Matrix: A Randomized, Controlled Clinical Tria.
Brief Title: Implant Placement and Simultaneous Soft Tissue Grafting With Single or Double Layers of Acellular Dermal Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12.0330
Record Dates: First submitted 2013-07-07; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Clinical Efficacy
Keywords: allograft; acellular dermal matrix; Alloderm
MeSH Terms: interventions — Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- one layer allograft (Active Comparator): One layer allograft as a positive control
  Interventions: Procedure: One layer allograft
- Two layer allograft (Experimental): Two layer allograft as the test group.
  Interventions: Procedure: Two layer allograft

INTERVENTIONS:
Procedure: One layer allograft — The acellular dermal matrix was placed on the facial surface.
  Other Names: One layer of acellular dermal matrix (Alloderm).
  Arms: one layer allograft
Procedure: Two layer allograft — The acellular dermal matrix was placed on the facial surface.
  Other Names: Two layers of acellular dermal matrix (Alloderm).
  Arms: Two layer allograft

SUMMARY:
The purpose of this study is to compare the effect on soft tissue thickness of placing either a single or double layer of acellular dermal matrix simultaneous with dental implant placement. The hypothesis is that 2 layers of acellular dermal matrix will produce thicker tissues that one layer.

DETAILED DESCRIPTION:
Patients must be greater that 18 years old, not pregnant, and have an edentulous space with a tooth on each side that is treatment planned to receive a dental implant. The primary outcome measure is soft tissue thickness.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria were;

1. one edentulous site bordered by 2 teeth in the maxilla or mandible from first molar to first molar treatment planned to receive an implant
2. at least 18 years of age
3. must sign the informed consent -

Exclusion Criteria: The exclusion criteria included:

1. uncontrolled diabetes, immune disease, or any systemic disease that significantly affects the periodontium
2. previous head and neck radiation
3. oral bisphosphonates for > 3 years or any IV bisphosphonates
4. smoking > 1/2 pack per day or other tobacco habits that might interfere with soft tissue healing
5. requirement for prophylactic antibiotics
6. allergies to any medication or material used in the study, or that would adversely affect study procedures
7. chemotherapy in the previous 12 months
8. psychological problems that would interfere with treatment
9. patients unable or unwilling to sign the informed consent
10. pregnancy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Soft tissue thickness. | 4 months
  Determining the soft tissue thickness using a tissue probe.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic, School of Dentistry, University of Louisville, Louisville, Kentucky, United States